CLINICAL TRIAL: NCT00852293
Title: The Connection Between Liver Disease and Chitinase Proteins
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Adar Tomer MD, Hadassah Hebrew University Medical Center
Other Study IDs: 481132-HMO-CTIL
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Liver Disease
Keywords: liver disease; Chitinase 3 like-1 protein
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests are taken to determin Chitinase 3 like-1 protein levels.

GROUPS / COHORTS (1):
- study group: Patients with liver disease followed at the liver unit at Hadassah Medical Center.
  Interventions: Other: A blood test

INTERVENTIONS:
Other: A blood test — A blood test of about 5ml of blood will be taken to determine Chitinase 3 like-1 protein levels.

SUMMARY:
Chitinase and chitinase like proteins are members of the 18-glycosyl-hydrolase family. Several reports have linked the chitinase 3 like 1 protein with colitis, asthma and liver disease.

This study aims to evaluate the correlation of chitinase 3 like 1 protein with clinical parameters such as disease severity, reaction to treatment, portal hypertension and prognosis.

DETAILED DESCRIPTION:
Chitin is a poly saccharide, abundant in insects, fungi, crustaceans and other organisms, but not in mammals. Chitinases and chitinase like proteins (which have the ability to bind chitin without enzymatic activity) are members of the 18-glycosyl-hydrolase family. Their function and importance are still not clearly understood. However, several reports have linked the chitinase 3 like 1 protein with colitis and asthma. Furthermore, Johansen et al have reported elevated levels of chitinase 3 like 1 protein in patients with liver disease, mainly those with alcoholic liver disease (ALD) and fibrosis. This report consisted of 51 patients with ALD ,but only 16 and 17 patients with fatty liver and viral hepatitis respectively.

This study aims to evaluate the correlation of chitinase 3 like 1 protein with clinical parameters such as disease severity, reaction to treatment, portal hypertension (when measured) and prognosis.

***Study design:

a. Subjects i.The study will include patients with liver disease followed at the liver unit, Hadassah Medical Center, Jerusalem. b. Planned number i.The study is planned to include 200 volunteers. c. Inclusion criteria i.Patients with liver disease followed at the liver unit at Hadassah Medical Center. ii.Patients who have given their informed consent for participation in the study. d. Exclusion criteria i.Age<18y. ii.Pregnancy iii.Patients with other conditions associated with elevated chitinase 3 like 1 protein (such as asthma and rheumatoid arthritis). e. Chitinase 3 like-1 protein levels will be measured by a commercially available kit (Human Chitinase 3-like 1 Quantikine ELISA Kit, catalogue number - DC3L1, Biotest LTD). f. Stopping/modifying criteria i.At subjects' request. g. Trial entry and enrollment i.A consecutive cohort will be recruited form amongst the patients followed at the liver unit in Hadassah medical center. Jerusalem Israel. ii.Consenting patients will have a blood test drawn for chitinase 3 like 1 protein levels. iii.Clinical details of each patient will be obtained form the liver unit. iv.In addition to the routine follow up at the liver unit, follow up will be performed at 1,2 and 5 years. h. Statistical considerations i.Subjects will be grouped according to their clinical properties (disease, treatment, severity, portal hypertension) ii.Chitinase 3 like 1 protein levels will be compared between each group. F. Informed consent i.Each subject will be enrolled and enter the study only after giving an informed consent. G. Adherence to study eligibility i.The study will be conducted in accordance with good clinical practice (GCP) guidelines, and the study protocol. H. Safeguarding of documents i.The privacy of the subjects and all confidentiality issues will be handled in accordance with applicable law and guidelines of the institution and the Helsinki Committee, the Israeli ministry of health, or the other appropriate regulatory authorities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver disease followed at the liver unit at Hadassah Medical Center.
* Patients who have given their informed consent for participation in the study

Exclusion Criteria:

* Age<18y.
* Pregnancy
* Patients with other conditions associated with elevated chitinase 3 like 1 protein (such as asthma and rheumatoid arthritis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include patients with liver disease followed at the liver unit, Hadassah Medical Center, Jerusalem Israel.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Comparison between Chitinase 3 like-1 protein levels and liver disease parameters including disease severity, portal hypertension, reaction to treatment and prognosis. | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Background] Kawada M, Hachiya Y, Arihiro A, Mizoguchi E. Role of mammalian chitinases in inflammatory conditions. Keio J Med. 2007 Mar;56(1):21-7. doi: 10.2302/kjm.56.21. PMID 17392594
- [Background] Chupp GL, Lee CG, Jarjour N, Shim YM, Holm CT, He S, Dziura JD, Reed J, Coyle AJ, Kiener P, Cullen M, Grandsaigne M, Dombret MC, Aubier M, Pretolani M, Elias JA. A chitinase-like protein in the lung and circulation of patients with severe asthma. N Engl J Med. 2007 Nov 15;357(20):2016-27. doi: 10.1056/NEJMoa073600. PMID 18003958
- [Background] Johansen JS, Christoffersen P, Moller S, Price PA, Henriksen JH, Garbarsch C, Bendtsen F. Serum YKL-40 is increased in patients with hepatic fibrosis. J Hepatol. 2000 Jun;32(6):911-20. doi: 10.1016/s0168-8278(00)80095-1. PMID 10898311